CLINICAL TRIAL: NCT04151407
Title: A Phase I , Multicenter, Open-Label, Single/Multiple Dose- Escalation Study of Recombinant Humanized Anti-VEGF Monoclonal Antibody Injection in Patients With Diabetic Macular Edema(DME)
Brief Title: The Study of Drug 601 in Patients With Diabetic Macular Edema (DME)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-601-DME-I-01
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Macular Edema
Keywords: VEGF; DME; bevacizumab; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 601 dose level 1 treatment (Experimental): Recombinant humanized anti-VEGF monoclonal antibody, drug 601(0.375mg), Vitreous injection, injection once;
  Interventions: Drug: Drug 601
- 601 dose level 2 treatment (Experimental): Recombinant humanized anti-VEGF monoclonal antibody, drug 601(0.75mg), Vitreous injection, injection once
  Interventions: Drug: Drug 601
- 601 dose level 3 treatment (Experimental): Recombinant humanized anti-VEGF monoclonal antibody, drug 601(1.25mg), Vitreous injection, injection once
  Interventions: Drug: Drug 601
- 601 dose level 4 treatment (Experimental): Recombinant humanized anti-VEGF monoclonal antibody, drug 601(2.5mg), Vitreous injection, injection once;
  Interventions: Drug: Drug 601
- 601 dose level 5 treatment (Experimental): Recombinant humanized anti-VEGF monoclonal antibody, drug 601(3.75mg), Vitreous injection, injection once;
  Interventions: Drug: Drug 601
- 601 dose level 6 treatment (Experimental): Recombinant humanized anti-VEGF monoclonal antibody, drug 601(1.25mg), Vitreous injection, injection once every 4 weeks, three times continuously.
  Interventions: Drug: Drug 601
- 601 dose level 7 treatment (Experimental): Recombinant humanized anti-VEGF monoclonal antibody, drug 601(2.5mg), Vitreous injection, injection once every 4 weeks, three times continuously.
  Interventions: Drug: Drug 601

INTERVENTIONS:
Drug: Drug 601 — Drug is a kind of recombinant anti-VEGF humanized monoclonal antibody injection.

SUMMARY:
Observe the safety and tolerability of the single and multiple doses of 601 in DME patients; study the pharmacokinetic characteristics of single and multiple doses of 601, Observe the Preliminary efficacy of 601 multiple injections with different doses in the treatment of patients with DME.

DETAILED DESCRIPTION:
According to the results of preclinical pharmacological research and clinical application of bevacizumab in ophthalmology Case, 601 will be developed as a drug candidate for the treatment of ocular diseases such as DME .Observe the safety and tolerability of the single and multiple doses of 601 in DME patients; study the pharmacokinetic characteristics of single and multiple doses of 601, Observe the Preliminary efficacy of 601 multiple injections with different doses in the treatment of patients with DME.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form and willing to be visited at the time specified in the trial
* Age >= 18 years and age =< 75 years
* Diagnosis of type 1 or type 2 diabetes
* Hemoglobin (HbA1c) value =< 11%
* The study eye must meet the following criteria

  * Diabetic macular edema with central fovea involvement and visual impairment in subjects;
  * Best corrected visual acuity letter score (ETDRS)>= 19 (i.e., 20/400 or better) and <= 73 (i.e., 20/40 or worse)in the study eye;
  * CRT ≥ 275 μm;
  * No optometric media opacity and pupil shrinkage.
* Best corrected visual acuity letter score (ETDRS) > =24 (i.e., 20/320 or better)in the fellow eyes

Exclusion Criteria:

* Any eye has active ocular infections (e.g.,blepharitis, keratitis, scleritis, conjunctivitis);
* The study eye has proliferative diabetic retinopathy (PDR), except for the PDR with regression after panretinal photocoagulation, and Inactive, fibrotic PDR
* History of vitreous hemorrhage in the study eye within 2 months before screening
* Structural retinal damage with fovea in the study eye (e.g. retinal pigment epithelium(RPE) atrophy, retinal fibrosis, laser scarring, dense hard exudation), or researchers believe that the study eye has other retinal damage that may hinder visual improvement after macular edema subsides
* In addition to diabetic retinopathy, there are other causes of macular edema or visual changes in the study eye.

Ophthalmic conditions (e.g.,retinal vein occlusion (RVO) Choroidal neovascularization, retinal detachment, macular hole, retinal traction in macular region, epiretinal membrane, etc.)

* Iris neovascularization in the study eye;
* Uncontrollable glaucoma in the study eye (defined as intraocular pressure after antiglaucoma medication>= 25 mm Hg), or glaucoma filtering surgery history;
* Researchers believe that cataract in the study eye may affect the judgement of examination or test results, or surgical treatment is required in 6 months following screening
* The study eye has no lens( except intraocular lens)
* History of Intraocular injection for corticosteroids (e.g. triamcinolone) at any time in the past 3 months, or corticosteroids injection around the eyes within one month before screening
* History of vitrectomy in the studyeye
* History of panretinal photocoagulation in the study eye in the past 6 months before screening; or panretinal photocoagulation may be required following screening
* Study eye have received more than two local/grid retinal photocoagulation treatments, or history of local/grid retinal photocoagulation treatments in the study eye in the past 3 months before screening
* History of anti-VEGF drugs treatments(e.g. Abercept, Pigatani Sodium, Razumab, Bevacizumab, etc.) in any eye or system within 3 months before screening;
* History of any intraocular surgery (e.g. cataract surgery, YAG posterior capsulotomy, etc) in the study eye within 3 months before screening;
* History of ophthalmic surgery involving macular areas (e.g. PDT, macular transposition) in the study eye, except for local/grid retinal photocoagulation

Any of the following general condition are present:

* Uncontrolled blood pressure control (defined as systolic blood pressure > 150 mmHg or diastolic pressure > 95 mmHg after antihypertensive medication
* The subjects is suffering from systemic infections and requiring oral, intramuscular or intravenous medication
* History of stroke, transient ischemic attack, myocardial infarction or acute congestive heart failure in the past 6 months before screening;
* Medicines with toxicity to the lens, retina or optic nerve (deferoxamine, chloroquine,hydroxychloroquine (chloroquine), tamoxifen and phenol etc.) is being used or may be used during the study period
* Diagnosed systemic immune diseases (e.g. ankylosing spondylitis and systemic lupus erythematosus etc.), or any uncontrolled clinical problem (e.g. AIDS, malignant tumors, active hepatitis, serious mental, neurological, cardiovascular, respiratory and other systemic diseases, etc.)
* History of allergy to fluorescein sodium and allergies to protein products for treatment or diagnosis, history of allergy to more than two drugs and/or non-drug factors, or suffering from allergic diseases now

Any of the following laboratory tests abnormalities:

* Diabetic patients with uncontrolled blood glucose (fasting blood glucose >= 8.8 mmol/L);
* Renal function impairment (Cr is 1.5 times higher than the upper limit of normal values in the local laboratory) Liver dysfunction (ALT or AST is 2 times higher than the upper limit of normal value in the local laboratory).
* Abnormal coagulation function (prothrombin time >= the upper limit of normal value for 3 seconds) and activated partial thromboplastin time >= the upper limit of normal value for 10 seconds)

Patients with childbearing age with any of the following conditions:

- Those who do not use effective contraceptive measures;

The following are not excluded:

1. Natural amenorrhea for more than 12 months, or natural amenorrhea for 6 months and the serum follicle-stimulating hormone level > 40 mIU/mL;
2. Bilateral ovariectomy with/without hysterectomy for more than 6 weeks;
3. Use acceptable contraceptive methods(Sterilization, hormone contraception,Intrauterine device, double barrier method)
4. Be able to use reliable contraceptives throughout the study period and stick to the end of the visit, (Unacceptable contraceptive methods include regular abstinence by calendar, ovulation, body temperature measurement, post-ovulation and fertilization in vitro);

   * Pregnancy and lactation women (pregnancy is defined as urinary pregnancy test positive in this study)
   * Participation in any other drug clinical trials (except vitamins and minerals) in the past 1 month before screening
   * Researchers think it needs to be ruled out.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
DLT | From Day 0 up to Day 28
  Incidence of dose-limiting toxicities up to the Day 28
MTD | From Day 0 up to Day 56/112.
  Maximum tolerated dose

SECONDARY OUTCOMES:
Cmax | From Day 0 up to 56/112 days
  The maximum blood concentration after 601 drug enters the bloodstream
t1/2 | From Day 0 up to 56/112 days
  The half-life of drug 601, the time required for the terminal phase 601 drug concentration to drop by half
AUC | From Day 0 up to 56/112 days
  Area under the concentration-time curve, reflect the characteristics of the exposure of 601 drug in the body.
Vd | From Day 0 up to 56/112 days
  The proportional constant between the amount of 601 drug in the body and the blood concentration when the 601 drug achieves the dynamic balance in the body
CL | From Day 0 up to 56/112 days
  Clearance rate of drug 601 from the central ventricle.
MRT | From Day 0 up to 56/112 days
  The average length of time that the 601 drug stays in the body.
λz | From Day 0 up to 56/112 days
  the ratio of the amount of elimination of 601 drug from the body per unit time to the total amount in the body
Biomarker | From Day 0 up to 56/112 days
  Detection of VEGF concentration
Immunogenicity | From Day 0 up to 56/112 days
  Development of Anti-drug antibodies (ADA) after IVT injection of 601

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Chinese PLA General Hospital of Central Theater., Wuhan, Hubei
  - JiangSu Province Hospital, Nanjing, Jiangsu
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No